CLINICAL TRIAL: NCT02694367
Title: MAP Kinase Signaling Pathways Through ERK and p-ERK Protein in Human Placenta of Women With Recurrent Miscarriage
Brief Title: Expression of EPK in Recurrent Miscarriage
Acronym: EPK-RM
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: ERK
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent Miscarriage
Keywords: genetic basis
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Recurrent miscarriage group: Women with previous history of RM, defined as two or more consecutive miscarriages
  Interventions: Other: Investigate the MAP kinase signaling pathways through ERK and p-ERK proteins
- Control group: Women with no history of RM
  Interventions: Other: Investigate the MAP kinase signaling pathways through ERK and p-ERK proteins

INTERVENTIONS:
Other: Investigate the MAP kinase signaling pathways through ERK and p-ERK proteins

SUMMARY:
The present study is based on hypotheses that some as yet unknown genetic factors may result in recurrent miscarriage (RM). Consequently, the main aim of this study was to gain new information about the underlying genetic causes of RM in the Egyptian population and to investigate the expression of ERK and p-ERK protein in human placenta and their corresponding tissue, to assess the significance of MAPK signal pathway in progression of recurrent miscarriage and PI3K-Akt Pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age less than 12 weeks.
2. no uterine abnormalities (examined by ultrasonography or hysterosonogram)
3. previous history of RM, defined as two or more consecutive miscarriages

Exclusion Criteria:

1. Gestational age 12 weeks or more.
2. Endocrine etiology like (thyroid dysfunction, and uncontrolled diabetes mellitus).
3. Antiphospholipid syndrome, inherited thrombophilias, alloimmune causes.
4. Uterine anatomic anomalies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women fulfilling the eligibility criteria had been tested and complete history and examination was done
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The levels of ERK and AKT in placenta | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No